CLINICAL TRIAL: NCT02512068
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Comparative Study and a Phase 3, Multicenter, Open-label, Long-term Study to Evaluate the Efficacy and Safety of SYR-472 When Orally Administered at a Dose of 25 mg Once Weekly in Patients With Type 2 Diabetes Mellitus Complicated by Severe Renal Impairment or End-stage Renal Disease
Brief Title: A Phase 3, Randomized, Double-blind, Parallel-group, Comparative Study and a Phase 3, Multicenter, Open-label, Long-term Study of SYR-472 (25 mg) in Patients With Type 2 Diabetes Mellitus Complicated by Severe Renal Impairment or End-stage Renal Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-472-3003; U1111-1172-1511 (Registry Identifier: WHO); JapicCTI-152970 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trelagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trelagliptin 25 mg (Experimental): Trelagliptin 25 mg tablet, orally, once weekly before breakfast for up to Week 52 (Period I + II)
  Interventions: Drug: Trelagliptin 25 mg
- Placebo and Trelagliptin 25 mg (Experimental): Placebo tablet, orally, once weekly before breakfast for up to Week 12 (Period I), followed by trelagliptin 25 mg tablet, orally, once weekly before breakfast for up to Week 52 (Period II)
  Interventions: Drug: Trelagliptin 25 mg; Drug: Placebo

INTERVENTIONS:
Drug: Trelagliptin 25 mg — Trelagliptin 25 mg Tablets
  Other Names: SYR-472
Drug: Placebo — Placebo Tablets
  Arms: Placebo and Trelagliptin 25 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of trelagliptin when administered at a dose of 25 mg once weekly using placebo as a control in patients with type 2 diabetes mellitus complicated by severe renal impairment or end-stage renal disease and inadequate glycemic control despite diet and/or exercise therapy (if given) or despite treatment with one antidiabetic drug in addition to diet and/or exercise therapy (if given); and to evaluate the long-term efficacy and safety of trelagliptin when administered at a dose of 25 mg once weekly to patients with type 2 diabetes mellitus complicated by severe renal impairment or end-stage renal disease.

DETAILED DESCRIPTION:
This is a phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group, comparative study (Treatment Period I) and a phase 3, multicenter, open-label, long-term study (Treatment Period II) to evaluate the efficacy and safety of trelagliptin when administered orally at a dose of 25 mg once weekly to patients with type 2 diabetes mellitus complicated by severe renal impairment or end-stage renal disease and inadequate glycemic control despite diet and/or exercise therapy (if given) or despite treatment with one antidiabetic drug in addition to diet and/or exercise therapy (if given).

ELIGIBILITY:
Inclusion Criteria:

1. The participant has a diagnosis of type 2 diabetes mellitus.
2. The participant has a fasting C-peptide value of 0.6 ng/mL or higher at the start of the screening period (Week -6) and Week -2 of the screening period.
3. The participant has a hemoglobin value of 10.0 g/dL or higher at the start of the screening period (Week -6) and Week -2 of the screening period.
4. The participant has a Haemoglobin A1c (HbA1c) value of 7.0% or higher but less than 10.0% at Week -2 of the screening period. For participants undergoing hemodialysis (with End-stage Renal Disease [ESRD]), those with a glycoalbumin value of 20% or higher could be enrolled even if their HbA1c value is below 7.0% at Week -2 of the screening period.
5. <HbA1c value of 7.0% or higher but less than 10.0% at Week -2 of the screening period> The participant has an HbA1c value difference between the start of the screening period (Week -6) and Week -2 of the screening period within 10.0%* of the HbA1c value at the start of the screening period (Week -6).

   <For participants undergoing hemodialysis (with ESRD), glycoalbumin value of 20% or higher and HbA1c value of below 7.0% at Week -2 of the screening period> The participant has a glycoalbumin difference between the start of the screening period (Week -6) and Week -2 of the screening period within 10.0%* of the glycoalbumin value at the start of the screening period (Week -6).

   *: rounded to one decimal place
6. The participant has been on a fixed diet and/or exercise therapy (if any) for at least 6 weeks prior to the start of the screening period (Week -6).
7. The participant meets any of the following:

   * The participant has not received any antidiabetic medications (including insulin preparations) from at least 6 weeks prior to the start of the screening period (Week -6).
   * The participant is being treated with one oral hypoglycemic drug* starting from at least 6 weeks prior to the start of the screening period (Week -6) at a fixed dose and regimen.

     *: any one of the following medications: mitiglinide calcium hydrate, repaglinide, acarbose, miglitol, or voglibose
   * The participant is being treated with one insulin preparation** starting from at least 6 weeks prior to the start of the screening period (Week -6) at a fixed dose and regimen (≤40 units/day) of the insulin preparation.

     * Any one of the following insulin monotherapies: mixed (short-acting or rapid-acting insulin containing no more than 30% volume), intermediate-acting, or long-acting soluble insulin preparations
8. The participant is not undergoing hemodialysis or peritoneal dialysis and has severe renal impairment [creatinine clearance (Ccr) <30 mL/min at the start of the screening period (Week -6)], or the participant is undergoing hemodialysis and has end-stage renal failure.
9. In the opinion of the investigator or sub-investigator, the initiation of hemodialysis or peritoneal dialysis at least within 12 weeks after starting the investigational product is not expected. [in cases where the participant is not undergoing hemodialysis or peritoneal dialysis (patients with severe renal impairment)]
10. The participant has been undergoing hemodialysis starting from at least 6 months prior to informed consent and, in the opinion of the investigator or sub-investigator, the participant is clinically stable. [in cases where the participant is undergoing hemodialysis (patient with end-stage renal failure)]
11. The participant is male or female and is aged 20 years or older at the time of informed consent.
12. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent until one month after the end of the study.
13. In the opinion of the investigator or sub-investigator, the participant is capable of understanding and complying with protocol requirements.
14. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.

Exclusion Criteria:

1. The participant has clinically evident hepatic impairment [e.g., aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2.5 times the upper limit of normal or total bilirubin of ≥2.0 mg/dL at the start of the screening period (Week -6) or at Week -2 of the screening period].
2. The participant has any serious cardiac diseases, cerebrovascular disorders, or serious pancreatic or hematological diseases (e.g., participants who require inpatient treatment or are hospitalized for treatment within 24 weeks prior to the start of the screening period).
3. The participant has severe ketosis, diabetic coma or precoma, type 1 diabetes, severe infection, before or after surgery, or severe external trauma.
4. The participant has hemoglobinopathy (sickle cell disease, thalassemia, etc.).
5. The participant experienced hypoglycemia (participants with a blood glucose value of ≤70 mg/dL or hypoglycemic symptoms) within 6 weeks prior to the start of the screening period or during the screening period (at least twice per week).
6. The participant has inadequately controlled hypertension.
7. For participants who are being treated with one antidiabetic agent, the participant was using at least two antidiabetic therapies on the day before 6 weeks prior to the start of the screening period (Week -6) (43 days prior to the start of the screening period).
8. The participant has malignancies.
9. The participant has a history of hypersensitivity or allergies to dipeptidyl peptidase 4 (DPP-4) inhibitors.
10. The participant has a history of gastrectomy or small intestinal resection.
11. The participant is a habitual drinker and consumes a daily average of more than 100 mL of alcohol.
12. The participant has a history of drug abuse (defined as the use of an illegal drug) or alcohol dependence.
13. The participant is required to take excluded medications during the study period.
14. The participant has previously received trelagliptin.
15. The participant received any other investigational products (including study drugs in a post-marketing clinical study) within 12 weeks prior to the start of the screening period.
16. The participant is participating in other clinical studies at the time of informed consent.
17. If female, the participant is pregnant or lactating or intending to become pregnant from the time of informed consent to within 1 month after the end of the study; or intending to donate ova during such time period.
18. The participant is an immediate family member of a study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
19. The participant is hospitalized during the screening period or is deemed as requiring hospitalization during the study period by the investigator or sub-investigator, unless the hospitalization is for short-term evaluations including complete health checkups or shunt (including shunt maintenance).
20. The participant is deemed ineligible for the study for any other reason by the investigator or sub-investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (49):
- Japan (49):
  - Anjo, Aichi-ken
  - Kasukabe, Aichi-ken
  - Nagoya, Aichi-ken
  - Toyohashi, Aichi-ken
  - Yatomi, Aichi-ken
  - Asahi, Chiba
  - Kisarazu, Chiba
  - Yotsukaidō, Chiba
  - Imabari, Ehime
  - Matsuyama, Ehime
  - Niihama, Ehime
  - Chikushino-shi, Fukuoka
  - Kasuga, Fukuoka
  - Kasuya-gun, Fukuoka
  - Kitakyushu, Fukuoka
  - Munakata, Fukuoka
  - Tajimi, Gifu
  - Takasaki, Gunma
  - Fukuyama, Hiroshima
  - Chitose, Hokkaido
  - Himeji, Hyōgo
  - Takarazuka, Hyōgo
  - Mito, Ibaragi
  - Sakai, Ibaragi
  - Fujisawa, Kanagawa
  - Kamakura, Kanagawa
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Sendai, Miyagi
  - Nakano, Nagano
  - Ueda, Nagano
  - Kasaoka, Okayama-ken
  - Setouchi, Okayama-ken
  - Fukaya, Saitama
  - Kumagaya, Saitama
  - Hamamatsu, Shizuoka
  - Yoshinogawa, Tokushima
  - Hachiōji, Tokyo
  - Itabashi-ku, Tokyo
  - Kunitachi, Tokyo
  - Uozu, Toyama
  - Shimonoseki, Yamaguchi
  - Ube, Yamaguchi
  - Akita
  - Kumamoto
  - Nagano
  - Niigata
  - Osaka
  - Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 41 investigative sites in Japan, from 7 August 2015 to 24 April 2018.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus complicated by severe renal impairment or end stage renal disease (ESRD) were enrolled in one of the two treatment groups: trelagliptin 25 milligram (mg) throughout Period I and II, Placebo in Period I followed by trelagliptin 25 mg in Period II.
Period: Overall Study
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Started | 55 | 52
Completed | 43 | 39
Not Completed | 12 | 13
Not completed — Pretreatment Event/Adverse Event | 8 | 6
Not completed — Major Protocol Deviation | 1 | 0
Not completed — Voluntary Withdrawal | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Reason Not Specified | 3 | 5

BASELINE CHARACTERISTICS:
Population: Randomized Set, Randomized set was defined as all participants who were randomized in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg | Total
Number analyzed (Participants) | 55 | 52 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (10.28) | 65.8 (10.46) | 65.8 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 38 | 39 | 77
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 55 | 52 | 107
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2]
  Kilogram (kg)/meter (m)^2 | 24.41 (3.525) | 24.97 (4.017) | 24.68 (3.765)
Duration of Diabetes [Mean (Standard Deviation); unit: Months] — Mean duration between start of study and first time of diagnosis of type 2 diabetes mellitus was reported.
  Months | 239.7 (116.80) | 219.3 (106.35) | 229.8 (111.79)
Exercise Program [Count of Participants; unit: Participants] — Participants with exercise program were indicated "Yes", and those with no exercise program were indicated "No".
  Participants
    Yes | 13 | 12 | 25
    No | 42 | 40 | 82
Undergoing Hemodialysis [Count of Participants; unit: Participants] — Participants with undergoing hemodialysis were indicated "Yes", and those with no undergoing hemodialysis were indicated "No".
  Participants
    Yes (End Stage Renal Disease) | 40 | 39 | 79
    No (Severe Renal Impairment) | 15 | 13 | 28
Antidiabetic Drug at the start of the screening period (Week -6) [Count of Participants; unit: Participants] — Participants with antidiabetic drug at the start of the screening period were indicated "Yes", and those with no antidiabetic drug were indicated "No".
  Participants
    Yes | 35 | 33 | 68
    No | 20 | 19 | 39
Antidiabetic Drug at the start of the screening period (Week -6): Rapid-acting Insulin Secretagogue [Count of Participants; unit: Participants] — Participants with rapid-acting insulin secretagogue at the start of the screening period were indicated "Yes", and those with no rapid-acting insulin secretagogue were indicated "No".
  Participants
    Yes | 9 | 8 | 17
    No | 46 | 44 | 90
Antidiabetic Drug at the start of the screening period (Week -6): Mitiglinide Calcium Hydrate [Count of Participants; unit: Participants] — The number of participants with mitiglinide calcium hydrate at the start of the screening period was reported.
  Participants | 5 | 3 | 8
Antidiabetic Drug at the start of the screening period (Week -6): Repaglinide [Count of Participants; unit: Participants] — The number of participants with repaglinide at the start of the screening period was reported.
  Participants | 4 | 5 | 9
Antidiabetic Drug at the start of the screening period (Week -6): α-Glucosidase Inhibitor [Count of Participants; unit: Participants] — Participants with α-glucosidase inhibitor at the start of the screening period were indicated "Yes", and those with no α-glucosidase inhibitor were indicated "No".
  Participants
    Yes | 8 | 12 | 20
    No | 47 | 40 | 87
Antidiabetic Drug at the start of the screening period (Week -6): Acarbose [Count of Participants; unit: Participants] — The number of participants with acarbose at the start of the screening period was reported.
  Participants | 0 | 2 | 2
Antidiabetic Drug at the start of the screening period (Week -6): Miglitol [Count of Participants; unit: Participants] — The number of participants with miglitol at the start of the screening period was reported.
  Participants | 3 | 2 | 5
Antidiabetic Drug at the start of the screening period (Week -6): Voglibose [Count of Participants; unit: Participants] — The number of participants with voglibose at the start of the screening period was reported.
  Participants | 5 | 8 | 13
Antidiabetic Drug at the start of the screening period (Week -6): Insulin Preparation [Count of Participants; unit: Participants] — Participants with insulin preparation at the start of the screening period were indicated "Yes", and those with no insulin preparation were indicated "No".
  Participants
    Yes | 18 | 13 | 31
    No | 37 | 39 | 76
Antidiabetic Drug at the start of the screening period (Week -6): Type of Insulin Preparation [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 17 | 12 | 29
    Pre-Mixed | 8 | 5 | 13
    Long-Acting | 9 | 7 | 16
Creatinine Clearance [Mean (Standard Deviation); unit: Milliliter (mL)/ minute (min)] | 10.7 (8.32) | 11.3 (8.29) | 11.0 (8.27)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 8.3 (7.28) | 8.7 (8.00) | 8.5 (7.61)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 7.57 (0.849) | 7.74 (1.049) | 7.65 (0.951)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: Milligram (mg)/deciliter (dL)] | 143.1 (32.58) | 151.1 (39.30) | 147.0 (36.05)
Glycoalbumin [Mean (Standard Deviation); unit: Percent] | 23.21 (4.091) | 24.29 (4.565) | 23.74 (4.341)
Fasting C-Peptide [Mean (Standard Deviation); unit: Nanogram (ng)/mL] | 7.07 (5.481) | 7.41 (4.580) | 7.23 (5.042)
Fasting Glucagon [Mean (Standard Deviation); unit: Picogram (pg)/mL] | 177.4 (55.40) | 165.7 (38.13) | 171.7 (47.93)
Dipeptidyl-Peptidase-4 (DPP-4) Activity [Mean (Standard Deviation); unit: Nanomole(nmol)/min/mL] — DPP-4 is an enzyme which degrades the hormone called glucagon-like peptide-1 (GLP-1) which stimulates insulin secretion when blood sugar value is high. The higher value indicates the higher enzyme activity.
  Nanomole(nmol)/min/mL | 8.4745 (1.98793) | 8.4200 (2.04675) | 8.4478 (2.00754)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at the End of Treatment Period I
Time Frame: Baseline (Week 0) and end of Treatment Period I (Up to Week 12)
Population: Full Analysis Set: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Percent HbA1c
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Number analyzed (Participants) | 55 | 52
Percent HbA1c | -0.71 (0.087) | 0.01 (0.089)
Statistical Analysis 1: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Test type: Superiority; p < 0.0001, ANCOVA; Least square (LS) mean difference = -0.72, 95% CI 2-sided [-0.966 to -0.473], Standard Error of Mean 0.124

2. Primary Outcome: Number of Participants Who Had One or More Treatment Emergent Adverse Event (TEAE) Before the Start of Study Drug Administration in Treatment Period II
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a drug (including the study drug). It does not necessarily have to have a causal relationship with this treatment (including the study drug). An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug (including the study drug), whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. Reported data is the number of participants reporting one or more TEAEs that occurred before the start of Treatment Period II in each group.
Time Frame: Up to Week 12
Population: Safety Analysis Set: The safety analysis set was defined as all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Number analyzed (Participants) | 55 | 52
Participants | 40 | 32

3. Primary Outcome: Number of Participants Who Had One or More TEAE Occurred After 1st Dose of Trelagliptin 25 mg Tablet
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a drug (including the study drug). It does not necessarily have to have a causal relationship with this treatment (including the study drug). An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug (including the study drug), whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. As to collect the safety data of long-term treatment with the active drug widely, the number of participants reporting one or more TEAEs that occurred after 1st dose of trelagliptin 25 mg, that is events in Period I and II for "Trelagliptin 25 mg" group and events in Period II for "Placebo and Trelagliptin 25 mg" group, was analyzed.
Time Frame: Up to Week 54
Population: Safety Analysis Set: The safety analysis set was defined as all participants who received at least one dose of the study drug. Number analyzed is the number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Number analyzed (Participants) | 55 | 48
Participants | 54 | 48

4. Secondary Outcome: Changes From Baseline in HbA1c
Description: Reported data was the change from baseline in HbA1c at each time point.
Time Frame: Baseline (Week 0) and Week 2, 4, 8, 12, and End of Treatment Period I (up to Week 12) and Period II (up to Week 52)
Population: Full Analysis Set: All randomized participants who received at least one dose of study drug. The analyzed numbers for each arm were participants who were evaluable for this outcome measure at the given time point.
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Number analyzed (Participants) | 55 | 52
Percent HbA1c
  At Week 2 | -0.24 (0.274) | 0.05 (0.260)
  At Week 4: number analyzed (Participants) | 55 | 51
  At Week 4 | -0.46 (0.370) | 0.02 (0.362)
  At Week 8: number analyzed (Participants) | 53 | 48
  At Week 8 | -0.64 (0.556) | -0.05 (0.530)
  At Week 12: number analyzed (Participants) | 49 | 48
  At Week 12 | -0.73 (0.576) | 0.03 (0.740)
  At the End of Treatment Period I | -0.70 (0.555) | 0.00 (0.731)
  At the End of Treatment Period II: number analyzed (Participants) | 55 | 48
  At the End of Treatment Period II | -0.76 (0.824) | -0.74 (0.843)
Statistical Analysis 1: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in HbA1c at Week 2 was compared between the treatment groups; Test type: Other; Point estimate = -0.28, 95% CI 2-sided [-0.385 to -0.180]
Statistical Analysis 2: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in HbA1c at Week 4 was compared between the treatment groups; Test type: Other; Point estimate = -0.48, 95% CI 2-sided [-0.621 to -0.338]
Statistical Analysis 3: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in HbA1c at Week 8 was compared between the treatment groups; Test type: Other; Point estimate = -0.58, 95% CI 2-sided [-0.797 to -0.367]
Statistical Analysis 4: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in HbA1c at Week 12 was compared between the treatment groups; Test type: Other; Point estimate = -0.71, 95% CI 2-sided [-0.975 to -0.441]
Statistical Analysis 5: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in HbA1c at End of Treatment Period I was compared between the treatment groups; Test type: Other; Point estimate = -0.70, 95% CI 2-sided [-0.948 to -0.452]

5. Secondary Outcome: Number of Participants Achieving <6.0%, <7.0%, and <8.0% HbA1c at the End of Treatment Period I and Period II
Time Frame: At the end of Treatment Period I (Up to Week 12) and Period II (Up to Week 52)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Number analyzed (Participants) | 55 | 52
Participants
  HbA1c <6.0% at the End of Treatment Period I: number analyzed (Participants) | 53 | 50
  HbA1c <6.0% at the End of Treatment Period I | 3 | 2
  HbA1c <6.0% at the End of Treatment Period II: number analyzed (Participants) | 53 | 46
  HbA1c <6.0% at the End of Treatment Period II | 7 | 8
  HbA1c <7.0% at the End of Treatment Period I: number analyzed (Participants) | 44 | 41
  HbA1c <7.0% at the End of Treatment Period I | 22 | 7
  HbA1c <7.0% at the End of Treatment Period II: number analyzed (Participants) | 44 | 37
  HbA1c <7.0% at the End of Treatment Period II | 22 | 18
  HbA1c <8.0% at the End of Treatment Period I: number analyzed (Participants) | 15 | 19
  HbA1c <8.0% at the End of Treatment Period I | 10 | 5
  HbA1c <8.0% at the End of Treatment Period II: number analyzed (Participants) | 15 | 15
  HbA1c <8.0% at the End of Treatment Period II | 11 | 8
Statistical Analysis 1: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; The data of participants achieving <6.0% at the end of Treatment Period I were compared between the treatment groups; Test type: Other; Point estimate = 1.7, 95% CI 2-sided [-6.598 to 9.919]
Statistical Analysis 2: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; The data of participants achieving <7.0% at the end of Treatment Period I were compared between the treatment groups; Test type: Other; Point estimate = 32.9, 95% CI 2-sided [14.194 to 51.660]
Statistical Analysis 3: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; The data of participants achieving <8.0% at the end of Treatment Period I were compared between the treatment groups; Test type: Other; Point estimate = 45.6, 95% CI 2-sided [15.528 to 75.700]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Reported data was the change from baseline in fasting plasma glucose at each time point.
Time Frame: Baseline (Week 0) and Week 2, 4, 8, 12, and End of Treatment Period I (up to Week 12) and Period II (up to Week 52)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Number analyzed (Participants) | 55 | 52
mg/dL
  At Week 2 | -12.9 (22.67) | 2.3 (20.78)
  At Week 4: number analyzed (Participants) | 55 | 51
  At Week 4 | -11.3 (31.25) | -2.6 (32.49)
  At Week 8: number analyzed (Participants) | 53 | 48
  At Week 8 | -12.7 (25.56) | -4.3 (27.28)
  At Week 12: number analyzed (Participants) | 49 | 48
  At Week 12 | -15.9 (31.95) | -0.3 (24.86)
  At the End of Treatment Period I | -14.8 (31.51) | 0.8 (25.50)
  At the End of Treatment Period II: number analyzed (Participants) | 55 | 48
  At the End of Treatment Period II | -14.3 (37.48) | -7.3 (34.31)
Statistical Analysis 1: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in fasting plasma glucose at Week 2 was compared between the treatment groups; Test type: Other; Point estimate = -15.2, 95% CI 2-sided [-23.59 to -6.88]
Statistical Analysis 2: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in fasting plasma glucose at Week 4 was compared between the treatment groups; Test type: Other; Point estimate = -8.7, 95% CI 2-sided [-20.98 to 3.58]
Statistical Analysis 3: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in fasting plasma glucose at Week 8 was compared between the treatment groups; Test type: Other; Point estimate = -8.3, 95% CI 2-sided [-18.76 to 2.11]
Statistical Analysis 4: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in fasting plasma glucose at Week 12 was compared between the treatment groups; Test type: Other; Point estimate = -15.6, 95% CI 2-sided [-27.14 to -4.03]
Statistical Analysis 5: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in fasting plasma glucose at End of Treatment Period I was compared between the treatment groups; Test type: Other; Point estimate = -15.6, 95% CI 2-sided [-26.67 to -4.62]

7. Secondary Outcome: Change From Baseline in Glycoalbumin
Description: Reported data was the change from baseline in glycoalbumin at each time point.
Time Frame: Baseline (Week 0) and Week 2, 4, 8, 12, and End of Treatment Period I (up to Week 12) and Period II (up to Week 52)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Number analyzed (Participants) | 55 | 52
Percent
  At Week 2 | -1.67 (1.137) | 0.10 (1.059)
  At Week 4: number analyzed (Participants) | 55 | 51
  At Week 4 | -2.46 (1.534) | -0.01 (1.474)
  At Week 8: number analyzed (Participants) | 53 | 48
  At Week 8 | -2.69 (2.038) | -0.21 (2.033)
  At Week 12: number analyzed (Participants) | 49 | 48
  At Week 12 | -2.85 (2.523) | -0.27 (2.563)
  At the End of Treatment Period I | -2.81 (2.401) | -0.15 (2.537)
  At the End of Treatment Period II: number analyzed (Participants) | 55 | 48
  At the End of Treatment Period II | -3.12 (2.580) | -3.06 (2.604)
Statistical Analysis 1: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in glycoalbumin at Week 2 was compared between the treatment groups; Test type: Other; Point estimate = -1.76, 95% CI 2-sided [-2.184 to -1.340]
Statistical Analysis 2: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in glycoalbumin at Week 4 was compared between the treatment groups; Test type: Other; Point estimate = -2.45, 95% CI [-3.030 to -1.870]
Statistical Analysis 3: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in glycoalbumin at Week 8 was compared between the treatment groups; Test type: Other; Point estimate = -2.48, 95% CI 2-sided [-3.289 to -1.679]
Statistical Analysis 4: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in glycoalbumin at Week 12 was compared between the treatment groups; Test type: Other; Point estimate = -2.66, 95% CI 2-sided [-3.608 to -1.715]
Statistical Analysis 5: Comparison: Trelagliptin 25 mg vs Placebo and Trelagliptin 25 mg; Change from baseline in glycoalbumin at End of Treatment Period I was compared between the treatment groups; Test type: Other; Point estimate = -2.66, 95% CI 2-sided [-3.608 to -1.715]

8. Secondary Outcome: Numbers of Participants With TEAE Related to Vital Signs Before the Start of Study Drug Administration in Treatment Period II
Description: Number of participants with a vital sign-related TEAE classified under the System Organ Class of "investigations," was reported.
Time Frame: Up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Number analyzed (Participants) | 55 | 52
Participants | 1 | 2

9. Secondary Outcome: Number of Participants With Markedly Abnormal Values of 12-Lead Electrocardiogram (ECG) Parameters Before the Start of Study Drug Administration in Treatment Period II
Description: Here "QTcF" is corrected QT interval by Fridericia formula.
Time Frame: Up to Week 12
Population: Safety Analysis Set: The safety analysis set was defined as all participants who received at least one dose of the study drug. The analyzed numbers for each arm were participants who were evaluable for this outcome measure at the given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Number analyzed (Participants) | 55 | 51
Participants
  QTcF Interval >450 millisecond (msec) | 13 | 16
  QTcF Interval >480 msec | 3 | 5
  QTcF Interval >500 msec | 1 | 1

10. Secondary Outcome: Number of Participants With Markedly Abnormal Values of Clinical Laboratory Parameters Before the Start of Study Drug Administration in Treatment Period II
Description: Here "U/L" is Unit/Litter, and "ULN" is Upper Limit of Normal.
Time Frame: Up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
Number analyzed (Participants) | 55 | 52
Participants
  Amylase (U/L) >2×ULN | 4 | 1
  Lipase (U/L) >3×ULN | 1 | 3

ADVERSE EVENTS:
Time Frame: Up to Week 54
Description: Reported data were number of participants who occurred at least one AEs for each arm and not for each intervention (Placebo versus Trelagliptin 25 mg) because collection of data for each intervention were not planned at the start of this study. Total number of participants at risk for each arm were defined as the participants who occurred at least one dose of trelagliptin 25 mg tablet under Safety Analysis Set defined as all participants who received at least one dose of the study drug.
Arm/Group | Trelagliptin 25 mg | Placebo and Trelagliptin 25 mg
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/48
Serious Adverse Events (participants affected / at risk) | 23/55 | 16/48
Other Adverse Events (participants affected / at risk) | 48/55 | 39/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trelagliptin 25 mg (N=55) | Placebo and Trelagliptin 25 mg (N=48)
Angina pectoris (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 3 | 0
Diabetic retinopathy (Eye disorders) | 3 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Cholangitis infective (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 2 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 1 | 0
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1
Dementia with Lewy bodies (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1
Subclavian vein stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trelagliptin 25 mg (N=55) | Placebo and Trelagliptin 25 mg (N=48)
Diarrhoea (Gastrointestinal disorders) | 4 | 7
Vomiting (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 1 | 5
Dental caries (Gastrointestinal disorders) | 3 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 24 | 16
Influenza (Infections and infestations) | 0 | 4
Fall (Injury, poisoning and procedural complications) | 12 | 5
Contusion (Injury, poisoning and procedural complications) | 8 | 7
Procedural hypotension (Injury, poisoning and procedural complications) | 3 | 3
Shunt stenosis (Injury, poisoning and procedural complications) | 3 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 3 | 2
Blood pressure decreased (Investigations) | 4 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 12 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Headache (Nervous system disorders) | 3 | 4
Dizziness (Nervous system disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 5 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Hypertension (Vascular disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT02512068/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT02512068/SAP_001.pdf